CLINICAL TRIAL: NCT05914831
Title: Ultra-hypofractionated for Whole Breast Irradiation (WBI) Compared to Partial Breast Irradiation (PBI): A Single-Institution Prospective Phase 2 Trial
Brief Title: Ultra-hypofractionated for Whole Breast Irradiation (WBI) Compared to Partial Breast Irradiation (PBI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Institute of Vojvodina (Other Government)
Responsible Party: Principal Investigator, Marko Bojovic, Ass. MD, Oncology Institute of Vojvodina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS-dojka-SRB
Record Dates: First submitted 2023-06-08; First posted 2023-06-22 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer Female
Keywords: Ultra-hypofractionated radiotherapy; Partial breast irradiation; Breast radiotherapy toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Partial Breast Irradiation (Active Comparator)
  Interventions: Radiation: Ultra-fractionated PBI
- Whole Breast Irradiation (Experimental)
  Interventions: Radiation: Ultra-fractionated WBI

INTERVENTIONS:
Radiation: Ultra-fractionated WBI — An ultra-short course of radiotherapy with 26Gy in 5 fractions will be administered to the whole breast where the tumor was located.
  Arms: Whole Breast Irradiation
Radiation: Ultra-fractionated PBI — An ultra-short course of radiotherapy with 26Gy in 5 fractions will be administered to the part of the breast where the tumor was located.
  Arms: Partial Breast Irradiation

SUMMARY:
Female patients undergoing surgical treatment for early breast cancer and meeting the inclusion criteria for adjuvant breast radiotherapy were randomized into two groups. One group will receive adjuvant whole-breast radiotherapy in ultra-hypofractionated regimen of 26 Gy in 5 fractions. In contrast, the other group will receive partial breast irradiation with a dose of 26Gy in 5 fractions.

The study's objective is to compare the effects of both breast radiotherapy protocols in terms of locoregional disease control and survival and to compare the adverse effects of radiotherapy between the two protocols. To determine if there is a correlation between different parameters and the efficacy and degree of toxicity for both protocols.

DETAILED DESCRIPTION:
Radiation therapy should ideally start 6-8 weeks after breast-conserving surgery but no later than 12 weeks after the surgery.

If adjuvant chemotherapy has been administered, it is recommended to start radiation therapy three weeks after chemotherapy (optionally, it can be completed before beginning chemotherapy).

The radiation therapy procedure follows the existing clinical protocol for breast radiotherapy. For radiation therapy planning, the patient is positioned supine using immobilization devices (such as a wing board or similar) to ensure daily reproducibility within a range of 5 mm. The clinical target volume (CTV) is delineated according to the recommendations of the Danish Breast Cancer Cooperative Group (DBCG) and the European Society for Radiotherapy and Oncology (ESTRO).

A total dose of 26Gy in 5 fractions every working day using the Volumetric Modulated Arc Therapy (VMAT) technique. Daily portal images are obtained, and a breathing control protocol is applied based on clinical assessment (for left breast radiation therapy, active breath control is used - in deep inspiration or respiratory gating).

ELIGIBILITY:
Inclusion Criteria:

* Breast-conserving surgery
* Invasive ductal carcinoma
* Age ≥ 50
* Tumor size ≤ 3 cm
* R0 resection
* Unicentric/unifocal carcinoma or multifocal carcinoma within 2 cm of the primary neoplasm
* pN0 (sentinel lymph node biopsy or axillary lymph node dissection performed), N1mi
* Hormone receptor status - any
* Histological grade G1 or G2

Exclusion Criteria:

* Neoadjuvant systemic therapy
* TNBC (triple-negative breast cancer)
* Extensive intraductal component (EIC)
* Lymphovascular invasion (LVI)
* associated DCIS > 2.5 cm in size or high nuclear grade

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 1-6 months after RT
  Assessment of acute toxicity of radiotherapy in two radiotherapy regimens. Acute toxicity will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0
Late toxicity | 6-60 months after RT
  Assessment of late toxicity of radiotherapy in two radiotherapy regimens. Acute toxicity will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) scale version 5.0

SECONDARY OUTCOMES:
Local-regional control | 3, 5 and 10 years
  Any newly suspicious skin change/s or palpable lymph node in the irradiated area that is/are pathologically proved to be locoregional tumor recurrence.
Disease-free survival | 3, 5 and 10 years
  Disease-free survival refers to the time from adjuvant radiotherapy of breast cancer to clinically confirmed local recurrence, distant metastasis, second primary tumor diagnosis, or patient death.
Overall Survival | 3, 5 and 10 years
  Time from adjuvant radiotherapy to death.
Distant metastasis occurrence | 3, 5 and 10 years
  The time from adjuvant radiotherapy to the occurrence of distant metastasis.
Cosmetic outcome | at baseline, during the radiotherapy, immediately after radiotherapy termination and then in the first 2 years every 3 months, in the 4th and 5th year every 6 months and after 5 years once per year.
  The Harvard score for breast cosmesis (a 4-grade scale) will be used, which will be independently filled out by both patients and physicians.
QoL assessment | at baseline, during the radiotherapy, immediately after radiotherapy termination and then in the first 2 years every 3 months, in the 4th and 5th year every 6 months and after 5 years once per year.
  We will use the EORTC QLQ-BR23 questionnaire validated for the Serbian-speaking population to assess the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
The analyzed data from the study will be published in scientific journals. We are prepared to share our data for analysis with researchers from similar studies (previously registered on ClinicalTrials.gov) to compare our results.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The expected time for the publication of the first data is in 3 years (2026).
Access Criteria: Contact the researchers via email.